CLINICAL TRIAL: NCT03170141
Title: Immunogene-modified Antigen-specific T (IgT) Cells for the Treatment of Glioblastoma Multiforme
Brief Title: Immunogene-modified T (IgT) Cells Against Glioblastoma Multiforme
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17003
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma Multiforme of Brain; Brain Cancer
Keywords: CAR T; Gene Therapy; GBM; GD2; CD276; PD1
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with GBM will be treated with tumor targeting IgT cells including CAR-T cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antigen-specific IgT cells (Experimental): Patients will receive non-myeloablative chemotherapy consisting of fludarabine and cyclophosphamide, followed by intravenous infusion of autologous IgT cells. The tested IgT cell dosage ranges from 5×10^5 /kg to 5×10^6 /kg
  Interventions: Biological: Antigen-specific IgT cells

INTERVENTIONS:
Biological: Antigen-specific IgT cells — Tumor antigen-specific IgT cells are infused intravenously . Drug: cyclophosphamide 250 mg/m^2 d1-3; Drug: Fludarabine 25mg/m^2 d1-3

SUMMARY:
This study aims to treat patients who have been diagnosed with brain cancer glioblastoma multiforme (GBM) including diffuse intrinsic pontine glioma (DIPG) and diffuse midline glioma (DMG). The treatment combines two different approaches to fight cancer: immune modulators and antigen-specific T cells. Immune checkpoint antibodies have been tested on various tumors with good outcomes. GBM is known to express increased levels of certain antigens that can be targeted by T cells including chimeric antigen receptor-modified T (CAR-T) cells and tumor antigen specific cytotoxic lymphocytes (CTLs). In this study, the gene-modified T cells specific for GBM antigens will be combined with immune modulatory gene-modified dendritic cells (DCs) as individualized treatment regimens to treat patients.

DETAILED DESCRIPTION:
Background:

Glioblastoma multiforme (GBM) is the most dangerous and aggressive form of brain cancer. Chimeric antigen receptor (CAR)-modified T cells have been shown to mediate long-term durable remissions in recurrent or refractory hematopoietic malignancies, and thus the CAR-T therapy approach is also considered a promising treatment against GBM. Some surface antigens such as GD2 and CD56 have been targeted as potential GBM antigens. In addition, certain antigens are highly specific in GBM, such as epidermal growth factor receptor variant EGFRviii and metastasis related antigen CD44v6.

Tumor microenvironment is known to suppressive anti-cancer immune responses. Many immune checkpoint inhibitors have demonstrated marked anti-tumor activities. For example, CD276 is a member of the B7 family of immune checkpoint proteins, and CD276-specific CAR-T cell therapy have been considered a potential brain tumor microenvironment treatment. Besides immune checkpoint inhibitor antibodies, antigen-specific T cells modified with immune modulatory genes (IgT) such as genes encoding immune checkpoint inhibitors may be applied. Combination of tumor targeting and immune modulatory activities, the IgT cells could target both the tumor cells and the tumor microenvironment.

ELIGIBILITY:
Inclusion Criteria:

1. abilities to understand and the willingness to provide written informed consent;
2. patients are ≥ 6 and ≤ 70 years old;
3. recurrent glioblastoma or brain tumor patients with measurable tumors. Patients have received standard care of medication, such as gross total resection with concurrent radio-chemotherapy (~54 - 60 Gy, TMZ). Patients must either not be receiving dexamethasone or receiving ≤ 4 mg/day at the time of leukopheresis;
4. karnofsky performance score (KPS) ≥ 60;
5. life expectancy >3 months;
6. satisfactory bone marrow, liver and kidney functions as defined by the following: absolute neutrophile count ≥ 1500/mm^3; hemoglobin > 10 g/dL; platelets > 100000 /mm^3; Bilirubin < 1.5×ULN; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5×ULN; creatinine < 1.5×ULN;
7. peripheral blood absolute lymphocyte count must be above 0.8×10^9/L;
8. satisfactory heart functions;
9. patients must be willing to follow the instructions of doctors;
10. women of reproductive potential (between 15 and 49 years old) must have a negative pregnancy test within 7 days of study start. Male and female patients of reproductive potential must agree to use birth control during the study and 3 months post study.

Exclusion Criteria:

1. a prior history of gliadel implantation 4 weeks before this study start or currently receiving antibody based therapies;
2. HIV positive;
3. tuberculosis infection not under control;
4. history of autoimmune disease, or other diseases require long-term administration of steroids or immunosuppressive therapies;
5. history of allergic disease, or allergy to immune cells or study product excipients;
6. patients already enrolled in other immune cell clinical study;
7. patients, in the opinion of investigators, may not be eligible or not able to comply with the study.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of infusion of autologous IgT cells with cyclophosphamide and fludarabine as lymphodepleting chemotherapy in patients with recurrent glioblastoma using the NCI CTCAE V4.0 criteria. | 1 years
  incidents of treatment related adverse events as assessed by CTCAE V4.0.

SECONDARY OUTCOMES:
Treatment response rate of recurrent glioblastoma | 6 months
  Defined as the proportion of patients who achieved complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD).
Overall survival Rate | 2 years
  Percentage of participants with objective response as determined by the investigator based on Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1)
Progression-free survival rate | 2 years
  Progression-free Survival (PFS) as determined by the investigator based on RECIST v1.1
Persistence and proliferation of IgT cells in patients | 2 years
  IgT cell percentage in the peripheral blood by qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Z, Zhou J, Yang X, Liu Y, Zou C, Lv W, Chen C, Cheng KK, Chen T, Chang LJ, Wu D, Mao J. Safety and antitumor activity of GD2-Specific 4SCAR-T cells in patients with glioblastoma. Mol Cancer. 2023 Jan 9;22(1):3. doi: 10.1186/s12943-022-01711-9. PMID 36617554